CLINICAL TRIAL: NCT01721941
Title: A Phase I Dose Escalation Study of TH-302 Plus Doxorubicin Delivered by Trans-Arterial Chemoembolization (TACE) in Patients With Hepatocellular Carcinoma
Brief Title: TH-302 Plus Doxorubicin Delivered by Trans-Arterial Chemoembolization (TACE) in Patients With Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Scripps Clinic Cancer Center (Other)
Collaborators: Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH302 TACE
Record Dates: First submitted 2012-10-08; First posted 2012-11-06 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; HCC; liver cancer; hepatoma; TACE; transarterial chemoembolization; TH302
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase I dose level -1 (Experimental): TH-302 25mg; Doxorubicin 50mg
  Interventions: Drug: Phase I Dose level -1
- Phase I Dose level 1 (Experimental): TH-302 50mg; doxorubicin 50mg
  Interventions: Drug: Phase I dose level 1
- Phase I Dose level 2 (Experimental): TH-302 100mg; doxorubicin 50mg
  Interventions: Drug: Phase I Dose level 2
- Phase 1 Dose level 3 (Experimental): TH-302 150mg; Doxorubicin 50mg
  Interventions: Drug: Phase I Dose level 3

INTERVENTIONS:
Drug: Phase I Dose level -1 — The dose of TH-302 will be mixed with doxorubicin 50mg to use as the chemoembolization mixture for transarterial chemoembolization (TACE).
  Arms: Phase I dose level -1
Drug: Phase I dose level 1 — The dose of TH-302 will be mixed with doxorubicin 50mg to use as the chemoembolization mixture for transarterial chemoembolization (TACE).
  Arms: Phase I Dose level 1
Drug: Phase I Dose level 2 — The dose of TH-302 will be mixed with doxorubicin 50mg to use as the chemoembolization mixture for transarterial chemoembolization (TACE).
  Arms: Phase I Dose level 2
Drug: Phase I Dose level 3 — The dose of TH-302 will be mixed with doxorubicin 50mg to use as the chemoembolization mixture for transarterial chemoembolization (TACE).
  Arms: Phase 1 Dose level 3

SUMMARY:
The primary objective of this phase I dose escalation study is to determine the maximum tolerated dose of TH-302 when administered with doxorubicin via trans-arterial chemo-embolization (TACE) in patients with hepatocellular carcinoma (HCC) who are not transplant candidates and have unresectable disease. HCC is the second leading cause of worldwide cancer death and is generally incurable without liver transplant. TACE can convert about 40% of these patients to transplant candidates. Additionally, in non-transplant HCC patients, TACE confers statistical improvements in overall survival. Selective HCC arterial catheterization during TACE allows for the delivery of concentrated drugs to the liver tumor but the optimal TACE chemotherapy regimen has not yet been determined. TH-302 is a hypoxia inducible agent that can be activated in the hypoxic environment induced by TACE.

DETAILED DESCRIPTION:
Transarterial chemoembolization (TACE) is the major modality utilized for tumor downstaging for transplant and for local therapy in non-transplant patients. This procedure allows delivery of concentrated drugs to the tumor, followed by embolization that eliminates its blood supply creating an environment of hypoxia. The process induces tumor ischemia, while achieving a drug concentration in the tumor 10 to 25 times greater than can be achieved by infusion.

A hypoxic microenvironment is a characteristic of many solid tumors including hepatocellular cancer, further induced by TACE. The hypoxia-activated prodrug, TH-302, is designed to selectively physiologically target the hypoxic microenvironment. While doxorubicin and cisplatin have been used as the drugs in TACE among other agents, none have stood out as the optimal agent in targeting HCC. Because of the action of TH-302 in hypoxia, this agent has a mechanistic advantage as a agent in TACE.

The current study is designed to assess the potential therapeutic benefit of adding TH-302 to the standard doxorubicin based TACE regimen in patients with advanced hepatocellular carcinomas.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee
* Patients with hepatocellular carcinoma with either:

  1. liver limited disease who are not transplant candidates as they fall outside of Milan criteria, but may be eligible for transplant after successful downstaging with TACE
  2. liver limited disease who satisfy Milan criteria, but are at risk of falling out of Milan criteria before they receive a liver transplant
  3. non-transplantable HCC but with liver limited or metastatic disease that requires local TACE therapy
* Measurable disease by modified RECIST criteria (at least one target lesion outside of previous radiation fields)
* ECOG performance status of 2 or less
* Life expectancy of at least 3 months
* Childs-Pugh Class A or B
* HCC amenable to TACE
* Patent main portal vein (thrombosis of portal vein branch not exclusionary)
* Acceptable liver function:
* Bilirubin < 2 mg/dL
* AST (SGOT) and ALT (SGPT) < 5 x ULN is allowed
* Acceptable renal function:
* Serum creatinine < 1.5 ULN
* Acceptable hematologic status (without hematologic support for TACE #1):
* ANC > 500 cells/μL
* Platelet count > 50,000/μL

Exclusion Criteria:

* New York Heart Association (NYHA) Class III or IV, cardiac disease, myocardial infarction within 6 months prior to Day 1, unstable arrhythmia or symptomatic peripheral arterial vascular disease
* Known brain, leptomeningeal or epidural metastases (unless treated and well controlled for >=3 months)
* Previously treated malignancies, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years
* Severe chronic obstructive or other pulmonary disease with hypoxemia (requires supplementary oxygen, symptoms due to hypoxemia or oxygen saturation <90% by pulse oximetry after a 2 minute walk) or in the opinion of the investigator any physiological state likely to cause systemic or regional hypoxemia
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Sorafenib within the previous 4 weeks or the intention to initiate sorafenib while on study
* Poor liver function as indicated by serum bilirubin > 2 mg/dL, Child-Pugh Class C, severe coagulopathy (INR > 2) not correctable with vitamin K, or active hepatic encephalopathy
* Main portal vein occlusion
* Liver rupture or tumor penetration of liver capsule
* Tumor invasion of biliary system with biliary obstruction
* Severe cytopenias, including ANC < 500 cells/μL, Hemoglobin < 8 g/dL, or platelets < 50,000/μL
* Subjects who have exhibited allergic reactions to a structural compound, biological agent similar to TH-302
* Females who are pregnant or breast-feeding
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Unwillingness or inability to comply with the study protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of TH-302 use in TACE | 33 weeks
  Maximum tolerated dose (MTD) of TH-302 when co-administered with doxorubicin via TACE in patients with advanced hepatocellular cancer will be assessed with a Fibonacci (3+3) dose escalation design.

SECONDARY OUTCOMES:
Objective response rate | 12 months
  Assess overall response rate using standard RECIST criteria measured by triple phase CT or MRI at least 6 weeks post TACE administration

CONTACTS AND LOCATIONS:
Overall Officials: Darren S Sigal, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Clinic, La Jolla, California, United States